CLINICAL TRIAL: NCT00365378
Title: Study of Pilot Manufacturing Lot of HPV 16 Virus-Like Particle (VLP) Vaccine in the Prevention of HPV 16 Infection in 16- to 23-Year-Old Females
Brief Title: Study of Human Papillomavirus (HPV) 16 Vaccine in the Prevention of HPV 16 Infection in 16- to 23-Year-Old Females (V501-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-005; 2006_515
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2010-04-09 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: HPV 16 Infection
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): HPV 16 L1 VLP vaccine
  Interventions: Biological: Comparator: HPV 16 L1 Vaccine
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Comparator: Placebo

INTERVENTIONS:
Biological: Comparator: HPV 16 L1 Vaccine — A 0.5 intramuscular injection given at Day 1, Month 2, and Month 6
  Other Names: V501
  Arms: 1
Biological: Comparator: Placebo — A 0.5 intramuscular placebo injection given at Day 1, Month 2, and Month 6
  Arms: 2

SUMMARY:
Subjects received HPV 16 L1 VLP vaccine or placebo (1:1 ratio). Endpoints included efficacy, immunogenicity, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, unmarried females age 16 to 23 years with intact uteri
* Not pregnant at enrollment
* Agreed to use effective contraception through Month 7 of the study
* A lifetime history of 0 to 5 male partners with whom the subjects engaged in at least one episode of insertive intercourse

Exclusion Criteria:

* No prior history of Human Papillomavirus (HPV) vaccination
* No receipt of any other vaccination within 1 month prior to enrollment or plans to receive any other vaccination within 1 month prior to or after any dose of study vaccine
* No prior history of an abnormal Papanicolaou (Pap) test showing Squamous intraepithelial lesion (SIL) or biopsy showing Cervical intraepithelial neoplasia (CIN)

Ages: 16 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2409 (Actual)
Dates: Start 1999-09; Primary Completion 2004-03 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Mao C, Koutsky LA, Ault KA, Wheeler CM, Brown DR, Wiley DJ, Alvarez FB, Bautista OM, Jansen KU, Barr E. Efficacy of human papillomavirus-16 vaccine to prevent cervical intraepithelial neoplasia: a randomized controlled trial. Obstet Gynecol. 2006 Jan;107(1):18-27. doi: 10.1097/01.AOG.0000192397.41191.fb. PMID 16394035
- [Background] Koutsky LA, Ault KA, Wheeler CM, Brown DR, Barr E, Alvarez FB, Chiacchierini LM, Jansen KU; Proof of Principle Study Investigators. A controlled trial of a human papillomavirus type 16 vaccine. N Engl J Med. 2002 Nov 21;347(21):1645-51. doi: 10.1056/NEJMoa020586. PMID 12444178
- [Background] Paavonen J; Future II Study Group. Baseline demographic characteristics of subjects enrolled in international quadrivalent HPV (types 6/11/16/18) vaccine clinical trials. Curr Med Res Opin. 2008 Jun;24(6):1623-34. doi: 10.1185/03007990802068151. Epub 2008 Apr 23. PMID 18435868
- [Background] Barr E, Gause CK, Bautista OM, Railkar RA, Lupinacci LC, Insinga RP, Sings HL, Haupt RM. Impact of a prophylactic quadrivalent human papillomavirus (types 6, 11, 16, 18) L1 virus-like particle vaccine in a sexually active population of North American women. Am J Obstet Gynecol. 2008 Mar;198(3):261.e1-11. doi: 10.1016/j.ajog.2007.09.001. PMID 18313445
- [Background] Ault KA; Future II Study Group. Effect of prophylactic human papillomavirus L1 virus-like-particle vaccine on risk of cervical intraepithelial neoplasia grade 2, grade 3, and adenocarcinoma in situ: a combined analysis of four randomised clinical trials. Lancet. 2007 Jun 2;369(9576):1861-1868. doi: 10.1016/S0140-6736(07)60852-6. PMID 17544766
- [Background] Fraser C, Tomassini JE, Xi L, Golm G, Watson M, Giuliano AR, Barr E, Ault KA. Modeling the long-term antibody response of a human papillomavirus (HPV) virus-like particle (VLP) type 16 prophylactic vaccine. Vaccine. 2007 May 22;25(21):4324-33. doi: 10.1016/j.vaccine.2007.02.069. Epub 2007 Mar 12. PMID 17445955
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Wiley DJ, Masongsong EV, Lu S, Heather L S, Salem B, Giuliano AR, Ault KA, Haupt RM, Brown DR. Behavioral and sociodemographic risk factors for serological and DNA evidence of HPV6, 11, 16, 18 infections. Cancer Epidemiol. 2012 Jun;36(3):e183-9. doi: 10.1016/j.canep.2011.12.007. Epub 2012 Jan 25. PMID 22277329

RESULTS

PARTICIPANT FLOW:
Groups:
- HPV 16 L1 VLP (Group 1): The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time study subjects in Group 1 were vaccinated (at Day 1, Month 2, and Month 6) with HPV (Human Papillomavirus) 16 Virus-Like Particle (VLP) Vaccine.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the HPV 16 VLP Vaccine from completion of the Vaccination Period at Month 7 through Month 48. (The Month 7 visit was to be scheduled to occur no earlier than 3 weeks and no later than 7 weeks following the Month 6 visit.)
- Placebo (Group 2): The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time study subjects in Group 2 were vaccinated (at Day 1, Month 2, and Month 6) with placebo.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received placebo from completion of the Vaccination Period at Month 7 through Month 48. (The Month 7 visit was to be scheduled to occur no earlier than 3 weeks and no later than 7 weeks following the Month 6 visit.)
- Extension: This group includes 400 subjects who received Monovalent HPV 16 L1 VLP vaccine or placebo during the base study. This includes subjects who previously discontinued from the study.
Period: Vaccination (Day 1 to Month 7)
Arm/Group | HPV 16 L1 VLP (Group 1) | Placebo (Group 2) | Extension
Started | 1204 | 1205 | 0
Entered Vaccination Period | 1193 | 1198 | 0
Completed | 993 | 1038 | 0
Not Completed | 211 | 167 | 0
Not completed — Randomized Not Vaccinated | 11 | 7 | 0
Not completed — Adverse Event | 4 | 5 | 0
Not completed — Lost to Follow-up | 88 | 75 | 0
Not completed — Pregnancy | 19 | 14 | 0
Not completed — Protocol Violation | 22 | 13 | 0
Not completed — Withdrawal by Subject | 50 | 44 | 0
Not completed — Other | 17 | 9 | 0
Period: Follow-up (Month 7 Though Month 48)
Arm/Group | HPV 16 L1 VLP (Group 1) | Placebo (Group 2) | Extension
Started | 993 | 1038 | 0
Completed | 835 | 836 | 0
Not Completed | 158 | 202 | 0
Not completed — Moved | 6 | 5 | 0
Not completed — Lost to Follow-up | 67 | 69 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Withdrawal by Subject | 73 | 104 | 0
Not completed — Other | 11 | 21 | 0
Period: Extension
Arm/Group | HPV 16 L1 VLP (Group 1) | Placebo (Group 2) | Extension
Started | 0 | 0 | 400
Completed | 0 | 0 | 203
Not Completed | 0 | 0 | 197
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Moved | 0 | 0 | 8
Not completed — Lost to Follow-up | 0 | 0 | 57
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 98
Not completed — Other | 0 | 0 | 31

BASELINE CHARACTERISTICS:
Groups:
- HPV 16 L1 VLP (Group 1): The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time study subjects in Group 1 were vaccinated (at Day 1, Month 2, and Month 6) with HPV (Human Papillomavirus) 16 Virus-Like Particle (VLP) Vaccine.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the HPV 16 VLP Vaccine from completion of the Vaccination Period at Month 7 through Month 48.
- Placebo (Group 2): The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time study subjects in Group 2 were vaccinated (at Day 1, Month 2, and Month 6) with placebo.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received placebo from completion of the Vaccination Period at Month 7 through Month 48.
- Total: Total of all reporting groups
Arm/Group | HPV 16 L1 VLP (Group 1) | Placebo (Group 2) | Total
Number analyzed (Participants) | 1204 | 1205 | 2409
Age, Continuous [Mean (Full Range); unit: years] | 20.0 [16 to 25] | 20.1 [16 to 23] | 20.1 [16 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1204 | 1205 | 2409
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 69 | 73 | 142
  Black | 94 | 114 | 208
  Hispanic American | 89 | 93 | 182
  Native American | 9 | 14 | 23
  White | 918 | 889 | 1807
  Other | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Persistent HPV 16 Infection
Description: Cases of persistent infection were those with detection of HPV 16 by PCR (Polymerase chain reaction) on at least 2 consecutive visits at least 4 months apart; or detection of HPV 16 in a cervical biopsy specimen showing pathologic evidence of CIN1 (Cervical intraepithelial neoplasia), CIN2 or CIN3 together with HPV 16 detected at the visit immediately before or after the biopsy; or detection of HPV 16 on a subject's last visit.
Time Frame: Through Month 48
Population: Per-protocol population: subjects must have no major protocol violations, must be seronegative to HPV 16 at Day 1 and PCR (Polymerase chain reaction) negative to HPV 16 through Month 7, and must provide follow-up data after Month 7
Measure: Number; unit: Incidence per 100 person-years
Arm/Group | HPV 16 L1 VLP (Group 1) | Placebo (Group 2)
Number analyzed (Participants) | 755 | 750
Incidence per 100 person-years | 0.3 | 4.9
Statistical Analysis 1: Comparison: HPV 16 L1 VLP (Group 1) vs Placebo (Group 2); Test type: Superiority or Other; Vaccine Efficacy = 94.3, 95% CI [87.8 to 97.7] — Vaccine Efficacy (% relative risk reduction) Confidence Interval based on binomial tail probabilities and not from a dispersion parameter

2. Primary Outcome: Incidence of HPV 16-related CIN1, CIN2 or C1N3
Description: Cases of HPV 16-related CIN1, CIN2 or CIN3 are those with detection of HPV 16 in a cervical biopsy specimen showing pathologic evidence of CIN1, CIN2 or CIN3 together with HPV 16 detected at the visit immediately before or after the biopsy.
Time Frame: Through Month 48
Population: Per-protocol population: subjects must have no major protocol violations, must be seronegative to HPV 16 at Day 1 and PCR negative to HPV 16 through Month 7, and must provide follow-up data after Month 7
Measure: Number; unit: Incidence per 100 person-years
Arm/Group | HPV 16 L1 VLP (Group 1) | Placebo (Group 2)
Number analyzed (Participants) | 755 | 750
Incidence per 100 person-years | 0.0 | 1.0
Statistical Analysis 1: Comparison: HPV 16 L1 VLP (Group 1) vs Placebo (Group 2); Test type: Superiority or Other; Vaccine Efficacy = 100.0, 95% CI [84.0 to 100.0] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Serum Anti-HPV 16 Geometric Mean Titers
Description: The limit of detection of the assay was 6 mMU/ml. Samples with titer below the limit of detection were assigned a value of 3 for calculation of GMT and confidence interval. GMTs and confidence limits below the limit of detection are shown as "6.0".
Time Frame: Month 7
Population: Per-protocol population: subjects must have no major protocol violations, must be seronegative to HPV 16 at Day 1 and PCR negative to HPV 16 through Month 7, and must provide serology data at Month 7
Measure: Geometric Mean (95% Confidence Interval); unit: milliMerck units/ml (mMU/ml)
Arm/Group | HPV 16 L1 VLP (Group 1) | Placebo (Group 2)
Number analyzed (Participants) | 684 | 680
milliMerck units/ml (mMU/ml) | 1518.8 [1385.5 to 1665.0] | 6.0 [6.0 to 6.0]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from Day 1 until Month 7. No non-serious AEs were collected and no Vaccination Report Card (VRCs) were used in the extension study, therefore no data is entered for that group in the Other Adverse Events table.
Description: Subjects were observed for at least 20 minutes after each vaccination for any immediate reaction. Subjects were prompted to report temperatures and local (i.e., injection site) AEs for 5 days following each injection. Data on all other AEs were collected and recorded on the subject's vaccine report card for 14 days after each vaccination visit.
Groups:
- HPV 16 L1 VLP (Group 1); Placebo (Group 2): The number of subjects who actually received the vaccine material corresponding to the indicated vaccination group. There was one subject randomized to the HPV 16 L1 VLP vaccine group who received placebo and then discontinued study participation. There was 1 subject randomized to the placebo group who received one vaccination of HPV 16 L1 VLP vaccine and then discontinued study participation. These 2 subjects were included in the counts reported in the Adverse Event tables. There were 2 subjects randomized to the HPV 16 L1 VLP vaccine group and 2 subjects randomized to the placebo group and who received mixed vaccine material. These 4 subjects were not included in the counts reported in this table. Therefore, this table reports N=1191 (1193 minus 2) subjects vaccinated with HPV 16 L1 VLP vaccine and N=1196 (1198 minus 2) subjects vaccinated with placebo.
Arm/Group | HPV 16 L1 VLP (Group 1) | Placebo (Group 2) | Extension
Serious Adverse Events (participants affected / at risk) | 19/1191 | 20/1196 | 1/400
Other Adverse Events (participants affected / at risk) | 1025/1191 | 1013/1196 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HPV 16 L1 VLP (Group 1) (N=1191) | Placebo (Group 2) (N=1196) | Extension (N=400)
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radial nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2 | 0
Urinary bladder rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Limb deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Perineal laceration (Reproductive system and breast disorders) | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 0
Bulimia nervosa (Psychiatric disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0
Mania (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 2 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HPV 16 L1 VLP (Group 1) (N=1191) | Placebo (Group 2) (N=1196) | Extension (N=0)
Nausea (Gastrointestinal disorders) | 91 | 95 | 0
Fatigue (General disorders) | 59 | 64 | 0
Nasopharyngitis (Infections and infestations) | 85 | 88 | 0
Dizziness (Nervous system disorders) | 53 | 62 | 0
Headache (Nervous system disorders) | 499 | 495 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 68 | 65 | 0
Injection Site Erythema (General disorders) | 335 | 286 | 0
Injection Site Haematoma (General disorders) | 69 | 61 | 0
Injection Site Pain (General disorders) | 951 | 924 | 0
Injection Site Swelling (General disorders) | 288 | 211 | 0

LIMITATIONS AND CAVEATS:
Of note, the number of subjects reported in the results posting is slightly different than that specified in the publication by Koutsky, et al (2002). The data provided here is based on final data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.